CLINICAL TRIAL: NCT03334318
Title: PERL (Preventing Early Renal Loss in Diabetes) Continuous Glucose Monitoring (CGM) Study
Brief Title: PERL Continuous Glucose Monitoring (CGM) Study
Status: Completed | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); University of Minnesota (Other); University of Colorado, Denver (Other); University of Michigan (Other); Northwestern University Feinberg School of Medicine (Other); Albert Einstein College of Medicine (Other); Washington University School of Medicine (Other); University of Washington (Other); Providence Medical Research Center (Other)
Responsible Party: Principal Investigator, Alessandro Doria, Senior Investigator, Joslin Diabetes Center
Other Study IDs: 2018PG-T1D014
Record Dates: First submitted 2017-10-23; First posted 2017-11-07 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Time; Allopurinol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Allopurinol-treated: Participants in the PERL Clinical Trial (NCT02017171) randomized to allopurinol
  Interventions: Other: Mean blood glucose; Other: Blood glucose CV; Other: % time 70-180 mg/dL; Other: % time below 54 mg/dL; Other: % time above 180 mg/dL; Other: % time above 250 mg/dL; Other: MAGE (Mean amplitude of glucose excursions); Other: LBGI (Low Blood Glucose Index); Other: HBGI (High Blood Glucose Index); Drug: Allopurinol
- Placebo-treated: Participants in the PERL Clinical Trial (NCT02017171) randomized to placebo
  Interventions: Other: Mean blood glucose; Other: Blood glucose CV; Other: % time 70-180 mg/dL; Other: % time below 54 mg/dL; Other: % time above 180 mg/dL; Other: % time above 250 mg/dL; Other: MAGE (Mean amplitude of glucose excursions); Other: LBGI (Low Blood Glucose Index); Other: HBGI (High Blood Glucose Index); Drug: Placebo

INTERVENTIONS:
Other: Mean blood glucose — Mean of blood glucose values measures by continuous glucose monitoring from week 80 to week 164 of the PERL trial.
Other: Blood glucose CV — Coefficient of variation of blood glucose values measures by continuous glucose monitoring from week 80 to week 164 of the PERL trial.
Other: % time 70-180 mg/dL — Percent of time with blood glucose in the 70-180 mg/dL range as measured by continuous glucose monitoring from week 80 to week 164 of the PERL trial.
Other: % time below 54 mg/dL — Percent of time with blood glucose below 54 mg/dL as measured by continuous glucose monitoring from week 80 to week 164 of the PERL trial.
Other: % time above 180 mg/dL — Percent of time with blood glucose above 180 mg/dL as measured by continuous glucose monitoring from week 80 to week 164 of the PERL trial.
Other: % time above 250 mg/dL — Percent of time with blood glucose above 250 mg/dL as measured by continuous glucose monitoring from week 80 to week 164 of the PERL trial.
Other: MAGE (Mean amplitude of glucose excursions) — Mean amplitude of glucose excursions as measured by continuous glucose monitoring as measured by continuous glucose monitoring from week 80 to week 164 of the PERL trial.
Other: LBGI (Low Blood Glucose Index) — Low blood glucose index as measured by continuous glucose monitoring from week 80 to week 164 of the PERL trial.
Other: HBGI (High Blood Glucose Index) — High blood glucose index as measured by continuous glucose monitoring from week 80 to week 164 of the PERL trial.
Drug: Allopurinol — Oral allopurinol tablets administered in the PERL Clinical Trial
  Groups: Allopurinol-treated
Drug: Placebo — Oral placebo tablets administered in the PERL Clinical Trial
  Groups: Placebo-treated

SUMMARY:
Seven-point capillary profiles have shown that mean glucose correlates with both diabetic retinopathy and nephropathy risk. However, there remains great controversy as to whether the degree of variability around mean glucose may also contribute to these microvascular complications. The PERL trial (NCT02017171), testing whether treatment with allopurinol can slow down kidney function loss in type 1 diabetes, provides a unique opportunity to assess the role of glycemic variability in the progression of diabetic kidney disease in individuals who already have mild to moderate kidney disease. By applying Continuous Glucose Monitoring (CGM) in the PERL Study population, the investigators will be able to better understand how metrics of glycemia (mean, time above and below range, and various measures of variability) are associated with renal outcomes in the PERL population as a whole, but also in important subgroups (e.g., albuminuric vs. normoalbuminuric subjects with ongoing GFR decline, allopurinol vs. placebo arms). The nvestigators also aim to obtain precise information on the range of blood glucose corresponding to any given HbA1c value in this population since previous studies generally excluded patients with renal disease.

DETAILED DESCRIPTION:
Participants who consent to the study will have an Abbott Freestyle Libre Pro sensor placed on the back of their upper arm at their first PERL visit after this ancillary study has begun and at all subsequent PERL Visits. The sensor will be continuously worn by participants for 14 days. At the end of the 14 days, the sensor will be removed and mailed by the participant to the Coordinating center. Since subjects are at various stages of the PERL protocol, the number of remaining visits at which the CGM will be applied will vary among subjects.

STUDY AIMS

1. To assess the effect of glycemic variability, as measured by the coefficient of variation of CGM glucose (CV, the ratio of standard deviation and the mean of CGM glucose values), on the PERL renal functional endpoint (iohexol GFR at the end of study).
2. To assess the effect of other glycemic parameters measured by CGM (mean glucose, % time 70-180 mg/dL, % time below 54 mg/dL, % time below 70 mg/dL, % time above 180 mg/dL, % time above 250 mg/dL, mean amplitude of glucose excursions [MAGE], low blood glucose index [LBGI], high blood glucose index [HBGI]) on the PERL renal functional endpoint.
3. To assess the relationship between CGM-measured glycemic parameters and HbA1c at various levels of renal function.
4. To compare the effects of CGM metrics on the PERL renal endpoint and the corresponding effect of HbA1c.
5. To assess the effect of allopurinol treatment on all of the different glycemic metrics including HbA1c, CV, etc. and on their association with the PERL renal endpoint.

ELIGIBILITY:
Inclusion Criteria:

• Being an active participant in the PERL clinical trial

Exclusion Criteria:

* Having completed PERL Visit 16
* Pregnancy
* History of skin reactions in relation to the application of Abbott Freestyle Libre Pro

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of the PERL Clinical Trial
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
iGFR at the end of the PERL trial | Week 164 of the PERL trial
  Glomerular filtration rate (GFR) at the end of the PERL trial, measured by the plasma clearance of non-radioactive iohexol (iGFR) and adjusted for the iGFR at baseline.

SECONDARY OUTCOMES:
HbA1c at week 80 of the PERL trial | Week 80 of the PERL Trial
  Hba1c value at week 80 of the PERL trial
HbA1c at week 96 of the PERL trial | Week 96 of the PERL Trial
  Hba1c value at week 96 of the PERL trial
HbA1c at week 112 of the PERL trial | Week 112 of the PERL Trial
  Hba1c value at week 112 of the PERL trial
HbA1c at week 128 of the PERL trial | Week 128 of the PERL Trial
  Hba1c value at week 128 of the PERL trial
HbA1c at week 142 of the PERL trial | Week 142 of the PERL Trial
  Hba1c value at week 142 of the PERL trial
HbA1c at week 156 of the PERL trial | Week 156 of the PERL Trial
  Hba1c value at week 156 of the PERL trial
HbA1c at week 164 of the PERL trial | Week 164 of the PERL Trial
  Hba1c value at week 164 of the PERL trial
Mean blood glucose | From week 80 to week 164 of the PERL trial
  Mean of blood glucose values measured by continuous glucose monitoring
CV (coefficient of variation) of blood glucose | From week 80 to week 164 of the PERL trial
  Coefficient of variation of blood glucose values measured by continuous glucose monitoring
% time 70-180 mg/dL | From week 80 to week 164 of the PERL trial
  Percentage of time with blood glucose in the 70-180 mg/dL range (as measured by continuous glucose monitoring)
% time below 54 mg/dL | From week 80 to week 164 of the PERL trial
  Percentage of time with blood glucose below 54 mg/dL (as measured by continuous glucose monitoring)
% time above 180 mg/dL | From week 80 to week 164 of the PERL trial
  Percentage of time with blood glucose above 180 mg/dL (as measured by continuous glucose monitoring)
% time above 250 mg/dL | From week 80 to week 164 of the PERL trial
  Percentage of time with blood glucose above 250 mg/dL (as measured by continuous glucose monitoring)
MAGE (Mean amplitude of glucose excursions) | From week 80 to week 164 of the PERL trial
  Mean amplitude of glucose excursions as measured by continuous glucose monitoring
LBGI (Low blood glucose index) | From week 80 to week 164 of the PERL trial
  Low blood glucose index based on blood glucose values measured by continuous glucose monitoring
HBGI (High blood glucose index) | From week 80 to week 164 of the PERL trial
  High blood glucose index based on blood glucose values measured by continuous glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Doria, MD PhD MPH, Principal Investigator — Joslin Diabetes Center; Irl Hirsch, MD, Principal Investigator — University of Washington; Janet McGill, MD, Principal Investigator — Washington University, St. Louis, MO
Locations (19):
- United States (15):
  - Barbara Davis Center / University of Colorado Denver, Aurora, Colorado
  - Emory University - Grady Memorial Hospital, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Joslin Diabetes Center, Boston, Massachusetts
  - Brehm Center for Diabetes Research / University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - ICAHN School of Medicine at Mount Sinai, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Albert Einstein College of Medicine / Montefiore Medical Center, The Bronx, New York
  - UT Southwestern Dallas, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
- Canada (4):
  - Unversity of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - BC Diabetes, Vancouver, British Columbia
  - University of Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No